CLINICAL TRIAL: NCT05073939
Title: Effect of Oral Oxytocin of Brain and Behavioral Responses to Emotional Stimuli in Healthy Women
Brief Title: Effect of Oral Oxytocin on Women's Response to Emotional Stimuli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Principal Investigator, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-84
Record Dates: First submitted 2021-09-18; First posted 2021-10-12 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Oral Oxytocin; Emotional processing; Anxiety; Reward
MeSH Terms: conditions — Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Oxytocin (Experimental): Oxytocin orally (24 IU)
  Interventions: Drug: Oral Oxytocin
- Oral Placebo (Placebo Comparator): Placebo orally (identical ingredients, except the active agent)
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Oxytocin — Administration of oxytocin (24 international units) orally
  Other Names: Oxytocin Orally
  Arms: Oral Oxytocin
Drug: Oral Placebo — Administration of placebo orally
  Other Names: Placebo Orally
  Arms: Oral Placebo

SUMMARY:
The main aim of the study is to investigate whether orally administered oxytocin (24IU) could modulate females' neural and behavioral responses to affective stimuli including emotional faces and affective scenes.

DETAILED DESCRIPTION:
All subjects will complete a series of questionnaires firstly to control for possible pre-treatment confounders in terms of personality traits and mood: Beck Depression Inventory-II (BDI), Autism Spectrum Quotient (ASQ), Liebowitz Social Anxiety Scale (LSAS), State-Trait Anxiety Inventory (STAI), Childhood Trauma Questionnaire (CTQ), the Second Version of Social Responsiveness Scale(SRS-2), Positive and Negative Affect Schedule (PANAS). PANAS is administered before and after oral administration and after functional magnetic resonance imaging (fMRI) scanning. In the current double-blind, between-subject, placebo-controlled study 80 healthy female subjects will be recruited and receive oral administration either oxytocin (24IU) or placebo. Blood samples are collected twice before and 30 minutes after oral administration to assess the plasma OXT concentrations change. 45 minutes after oral administration subjects will be required to finish fMRI scanning including resting-state fMRI task, emotional face task (happy, fear, angry and neutral faces), affective scene task (NAPS, Nencki affective picture system, positive, neutral, and negative-valence scenes). After fMRI scanning, subjects will be required to rate valence, intensity, and arousal responses (Likert scale, 1-9 ratings) to the emotional and affective stimuli are presented during fMRI scanning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Head trauma
* Substance abuse
* Medication
* fMRI contraindications (e.g. metal implants)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes in blood oxytocin concentrations after oral oxytocin | Before and 30 minutes after treatment
  Changes in blood oxytocin concentrations will be assessed across two groups between baseline and 30 minutes after oral treatment administration.
Effects of oral oxytocin on neural responses to emotional faces assessed by emotional faces processing task fMRI | 45 minutes after treatment
  Comparison of neural activations between oral administration of oxytocin and placebo by means of treatment (oxytocin, placebo)× faces(happy, neutral, angry, fear) ANOVA and emotional face-specific post-hoc comparisons between the treatment groups.
Effects of oral oxytocin on neural responses to affective scenes assessed by affective scenes processing task fMRI | 45 minutes after treatment
  Comparison of neural activations as assessed by functional MRI on the whole-brain level between oral oxytocin and placebo by means of treatment (oxytocin, placebo) × scenes(neutral, positive, negative) ANOVA and scene-specific post-hoc comparisons between the treatment groups.
Effects of oral oxytocin on behavioral ratings of emotional faces stimuli | 45 minutes after treatment
  Differences in behavioral ratings of valence(1-9-point Likert scale, 1 means very negative,9 means very positive, 5 means neutral), intensity (1-9-point Likert scale, 1 means mild, 9 means strong), and arousal(1-9-point Likert scale, 1 means sleepy, 9 means alert) for emotional faces stimuli between oxytocin group and placebo group.
Effects of oral oxytocin on behavioral ratings of affective scenes stimuli | 45 minutes after treatment
  Differences in behavioral ratings of valence(1-9-point Likert scale, 1 means very negative,9 means very positive, 5 means neutral), intensity (1-9-point Likert scale, 1 means mild, 9 means strong), and arousal(1-9-point Likert scale, 1 means sleepy, 9 means alert) of affective scenes stimuli between oxytocin group and placebo group.

SECONDARY OUTCOMES:
The relationship between plasma oxytocin concentrations changes and neural responses to emotional faces stimuli | Before treatment to 150 minutes after treatment
  Correlation analysis between oral oxytocin-induced plasma oxytocin concentrations changes and oral oxytocin-induced neural responses/functional connectivity changes of emotional faces will be explored across two treatment groups.
The relationship between plasma oxytocin concentrations changes and neural responses to affective scenes stimuli | Before treatment to 150 minutes after treatment
  Correlation analysis between oral oxytocin-induced plasma oxytocin concentrations changes and oral oxytocin-induced neural responses/functional connectivity changes of affective scenes stimuli will be explored across two treatment groups.
The relationship between plasma oxytocin concentrations changes and behavioral responses to emotional faces stimuli | Before treatment to 150 minutes after treatment
  Correlation analysis between plasma oxytocin concentrations changes and post-scan behavioral ratings of emotional faces stimuli will be explored across two treatment groups.
The relationship between plasma oxytocin concentrations changes and behavioral responses to affective scenes stimuli | Before treatment to 150 minutes after treatment
  Correlation analysis between oral oxytocin-induced plasma oxytocin concentrations changes and post-scan behavioral ratings of affective scenes stimuli will be explored across two treatment groups.
Gender differences in plasma oxytocin concentrations changes | Before and 30 minutes after treatment
  Gender differences (male's data from ClinicalTrials.gov NCT04320706) in oral oxytocin-induced plasma oxytocin concentrations changes will be investigated.
Gender differences in neural response to emotional faces stimuli | 45 minutes after treatment
  Gender differences (male's data from ClinicalTrials.gov NCT04320706) in oral oxytocin-induced neural responses/functional connectivity to emotional faces stimuli will be investigated.
Gender differences in neural response to affective scenes stimuli | 45 minutes after treatment
  Gender differences (male's data from ClinicalTrials.gov NCT04320706) in oral oxytocin-induced neural responses/functional connectivity to affective scenes stimuli will be investigated.
Gender differences in behavioral responses to emotional faces stimuli | 45 minutes after treatment
  Gender differences (male's data from ClinicalTrials.gov NCT04320706) in oral oxytocin-induced post-scan behavioral responses to emotional faces stimuli will be investigated.
Gender differences in behavioral responses to affective scenes stimuli | 45 minutes after treatment
  Gender differences (male's data from ClinicalTrials.gov NCT04320706) in oral oxytocin-induced post-scan behavioral responses to affective scenes stimuli will be investigated.
Interaction effect between gender and treatment on plasma oxytocin concentrations changes | Before and 30 minutes after treatment
  The interaction effect between gender(male/female, male's data from ClinicalTrials.gov NCT04320706) and treatment(OXT/PLC) on plasma oxytocin concentrations changes will be investigated.
Interaction effect between gender and treatment on neural response to emotional faces stimuli | 45 minutes after treatment
  The interaction effect between gender(male/female, male's data from ClinicalTrials.gov NCT04320706) and treatment(OXT/PLC) on neural response/functional connectivity to emotional faces stimuli will be investigated.
Interaction effect between gender and treatment on neural response to affective scenes stimuli | 45 minutes after treatment
  The interaction effect between gender(male/female, male's data from ClinicalTrials.gov NCT04320706) and treatment(OXT/PLC) on neural response/functional connectivity to affective scenes stimuli will be investigated.
Interaction effect between gender and treatment on behavioral responses to emotional faces stimuli | 45 minutes after treatment
  The interaction effect between gender(male/female, male's data from ClinicalTrials.gov NCT04320706) and treatment(OXT/PLC) on post-scan behavioral ratings of emotional faces stimuli will be investigated.
Interaction effect between gender and treatment on behavioral responses to affective scenes stimuli | 45 minutes after treatment
  The interaction effect between gender(male/female, male's data from ClinicalTrials.gov NCT04320706) and treatment(OXT/PLC) on post-scan behavioral ratings of affective scenes stimuli will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China